CLINICAL TRIAL: NCT03667274
Title: Patient Outcome After Cardiac Double Valve Replacement at University Hospital Basel/ Switzerland
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-00553; ch18Grapow2
Record Dates: First submitted 2018-09-10; First posted 2018-09-12 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Cardiac Double Valve Replacement
Keywords: aortic valve replacement; mitral valve reconstruction; mitral valve replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cardiac valve surgery — cardiac double valve surgery (aortic and mitral valve)

SUMMARY:
To compare patient outcome data after cardiac double valve replacement (aortic and mitral valve) with patient outcome data after aortic valve replacement and mitral valve reconstruction

DETAILED DESCRIPTION:
To compare patient outcome data ( death, re-surgery, change in transvalvular gradient) after cardiac double valve replacement (aortic and mitral valve) with patient outcome data after aortic valve replacement and mitral valve reconstruction in patients with cardiac surgery at University Hospital Basel/ Switzerland since 2009.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing cardiac double valve surgery (aortic valve replacement, mitral valve replacement, mitral valve reconstruction) at University Hospital Basel/ Switzerland, starting 2009

Exclusion Criteria:

* denial of consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing cardiac double valve surgery (aortic valve replacement, mitral valve replacement, mitral valve reconstruction) at University Hospital Basel/ Switzerland, starting 2009
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
death | time from hospitalisation for cardiac valve surgery and following 12 months
  death after cardiac valve surgery
re-surgery | time from hospitalisation for cardiac valve surgery and following 12 months
  re-surgery after cardiac valve surgery
change in transvalvular gradient | time from hospitalisation for cardiac valve surgery and following 12 months
  change in transvalvular Gradient after cardiac valve surgery

CONTACTS AND LOCATIONS:
Overall Officials: Martin Grapow, Prof. Dr. MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- Herzchirurgie University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Egger ML, Gahl B, Koechlin L, Schomig L, Matt P, Reuthebuch O, Eckstein FS, Grapow MTR. Outcome of patients with double valve surgery between 2009 and 2018 at University Hospital Basel, Switzerland. J Cardiothorac Surg. 2022 Jun 13;17(1):152. doi: 10.1186/s13019-022-01904-9. PMID 35698233